CLINICAL TRIAL: NCT01799356
Title: Moxifloxacin Versus Ofloxacin Plus Metronidazole in Uncomplicated Pelvic Inflammatory Disease: Multicenter Randomized Controlled Trials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, Istanbul Sisli Etfal Training Research Hospital, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asicioglu03; treatment (Other: treatment pelvic inflammatuary disease); treatment uPID (Other: we aimed this study treatment uPID)
Record Dates: First submitted 2013-02-16; First posted 2013-02-26 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Treatment, moksifloksasin
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Moxifloxacin; Ofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- moxifloxacin Group (Active Comparator): Treatment at uPID with moxifloxacin
  Interventions: Drug: Moxifloxacin
- Ofloxacin Group (Placebo Comparator): Treatment at uPID with Ofloxacin plus metronidazole
  Interventions: Drug: Ofloxacin; Drug: Metronidazole

INTERVENTIONS:
Drug: Moxifloxacin — daily 400 mg moksifloksasin
  Other Names: new generetaion flouroquinolon antibiotics
  Arms: moxifloxacin Group
Drug: Ofloxacin — daily 800 mg oflaksasin plus 1000 mg metronidazol treatment
  Other Names: floroquinolon antibiotics
  Arms: Ofloxacin Group
Drug: Metronidazole — daily 1000 mg metronidazol plus 800 mg oflaksasin treatment for uPID
  Other Names: anaerobic antibiotics
  Arms: Ofloxacin Group

SUMMARY:
We aimed to compare efficacy and safety of combination therapy with oral ofloxacin, 400 mg twice daily, plus oral metronidazole, 500 mg twice daily, for 14 days, with moxifloxacin monotherapy, 400 mg once daily, for 14 days

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed uncomplicated PID
2. Patients age are between 14 with 45
3. Pelvic tenderness and vaginal discharge

Exclusion Criteria:

1. Urinary Tract Enfections
2. Tubo-ovarian abscess and complicated PID
3. Hıstory of antibiotics treatment
4. Other pelvic pain causes
5. Endometriosis
6. Delivery,abortion and surgery within last months

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1303 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clinically cure | 21 Days

SECONDARY OUTCOMES:
Microbiological cure | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Gungorduk, md, Study Chair — T.C.S.B. Kanıni Sultan Suleyman Training Hospital
Locations (4):
- Turkey (Türkiye) (4):
  - T.C.S.B. İstanbul Training Research Hospital, Samatya, Fatih
  - T.C.S.B. Kanuni Sultan Suleyman Training Hospital, Istanbul, Kucukcekmece
  - T.C.S.B Mardin Women and Children Hospital, Mardin, Mardin
  - T.C.S.B. Şişli Etfal Training Research Hospital, Şişli, Şişli

REFERENCES:
- [Result] Judlin P, Liao Q, Liu Z, Reimnitz P, Hampel B, Arvis P. Efficacy and safety of moxifloxacin in uncomplicated pelvic inflammatory disease: the MONALISA study. BJOG. 2010 Nov;117(12):1475-84. doi: 10.1111/j.1471-0528.2010.02687.x. Epub 2010 Aug 18. PMID 20716255
- [Result] Boothby M, Page J, Pryor R, Ross JD. A comparison of treatment outcomes for moxifloxacin versus ofloxacin/metronidazole for first-line treatment of uncomplicated non-gonococcal pelvic inflammatory disease. Int J STD AIDS. 2010 Mar;21(3):195-7. doi: 10.1258/ijsa.2009.009374. PMID 20215625
- [Derived] Savaris RF, Fuhrich DG, Maissiat J, Duarte RV, Ross J. Antibiotic therapy for pelvic inflammatory disease. Cochrane Database Syst Rev. 2020 Aug 20;8(8):CD010285. doi: 10.1002/14651858.CD010285.pub3. PMID 32820536